CLINICAL TRIAL: NCT03805204
Title: Anatomical Study About the Vascularization of the Ulna: Vascular and Mechanical Risk Factors Associated With Forearm Nonunion
Brief Title: Vascularity of the Ulna and Its Association With Forearm Nonunion
Acronym: Nonunion
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-CUB-2018-61
Record Dates: First submitted 2018-12-21; First posted 2019-01-15 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Forearm Fracture
MeSH Terms: interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Open reduction and internal fixation (ORIF) — ORIF with a forearm plate

SUMMARY:
Non-union after operative treatment of an ulnar fracture is very uncommon. There are severely disabling and challenging to treat. Multiple factors have been associated with the establishment of this non-union. Many non-unions are associated with soft tissue damage, fracture site vascularity, persistent instability, infection, and the surgical treatment technique. This study analysed the systemic conditions and local factors associated with the failure of bone fracture healing The aim of our study was to identify the risk factors for ulnar nonunion

DETAILED DESCRIPTION:
In the anatomical study we investigated the extraosseous and intraosseous blood supply in fourteen specimens from the Department of Human Anatomy. We correlated the areas with a low vascularity with the usual areas that patients have ulnar nonunion.

In the clinical study we retrospectively reviewed a cohort of ulnar fractures treated surgically with open reduction and internal fixation (ORIF), during a period of 10 years (2007-2016). We identified 211 ulnar fractures. All patients had a minimum follow-up of 1 year. We defined non-union if there was no radiological consolidation of the fracture after this period, and we classified them according to Weber classification. We assessed risk factors like: fracture site vascularity, surgical treatment technique, biological factors of the patient, and the fracture's mechanism. We correlated data and associated risk factors from the anatomical and the clinical studies.

Data were analysed using SPSS software system version 21. Multivariate regression analysis was performed to assess independent risk factors of ulnar non-union. Chi square test or Fisher exact test was used to compare categorical measurements. Statistical significance was considered as p less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adults from 18 to 90 years old
* Forearm ulnar nonunion

Exclusion Criteria:

* Children
* Other types of forearm fractures

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anatomical study: 14 upper extremities from the Department of Human Anatomy. Clinical study. Records about 211 ulnar fractures. We included only the fractures with the complication of ulnar nonunion.
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Avascular areas in anatomical study | 8 months
  The extraossea and intraossea vascularity of the forearms with Spalteholz dissection technique and Tompsett dissection technique will be described. The location, distribution and dimensions of the vessels and the areas without vascularity will be measured with a digital caliper (mm).
Epidemiological risk factors for ulnar nonunion | 8 months
  Epidemiological risks factor such as: smoke, heart problems, rheumatic disorders will be registered.
Biomechanical risk factors for ulnar nonunion | 8 months
  Biomechanical risk factors will be evaluated using the OTA/AO classification.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Lamas, Ph D, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
When we have the results we analyse the anatomical and clinical data and association with the differents risks factors in the Department of Statistics.

REFERENCES:
- [Background] Kloen P, Wiggers JK, Buijze GA. Treatment of diaphyseal non-unions of the ulna and radius. Arch Orthop Trauma Surg. 2010 Dec;130(12):1439-45. doi: 10.1007/s00402-010-1071-x. Epub 2010 Mar 9. PMID 20217106
- [Background] Kloen P, Buijze GA, Ring D. Management of forearm nonunions: current concepts. Strategies Trauma Limb Reconstr. 2012 Apr;7(1):1-11. doi: 10.1007/s11751-011-0125-0. Epub 2011 Nov 24. PMID 22113538
- [Background] Bartonicek J, Kozanek M, Jupiter JB. History of operative treatment of forearm diaphyseal fractures. J Hand Surg Am. 2014 Feb;39(2):335-42. doi: 10.1016/j.jhsa.2013.06.020. Epub 2013 Dec 11. PMID 24332651
- [Background] Hardy BT, Glowczewskie F Jr, Wright TW. Vascular anatomy of the proximal ulna. J Hand Surg Am. 2011 May;36(5):808-10. doi: 10.1016/j.jhsa.2011.02.011. Epub 2011 Apr 12. PMID 21489724
- [Background] Sheetz KK, Bishop AT, Berger RA. The arterial blood supply of the distal radius and ulna and its potential use in vascularized pedicled bone grafts. J Hand Surg Am. 1995 Nov;20(6):902-14. doi: 10.1016/S0363-5023(05)80136-4. PMID 8583061